CLINICAL TRIAL: NCT06663280
Title: Prospective Randomized Study to Prove a Positive Care Effect of the Digital Health Assistant ADELE Blood Pressure A0007 for Hypertension Patients
Brief Title: Positive Care Effect of the Digital Health Assistant ADELE Blood Pressure for Hypertension Patients
Acronym: A0007
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alma Phil Gmbh (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: APH01-2
Record Dates: First submitted 2024-10-19; First posted 2024-10-29 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Essential (Primary) Hypertension; Hypertensive Heart Disease With (Congestive) Heart Failure; Hypertensive Heart Disease Without (Congestive) Heart Failure; Other Secondary Hypertension; Secondary Hypertension, Unspecified; Syncope and Collapse; Dizziness and Giddiness
Keywords: hypertension; digital health; health assistant
MeSH Terms: conditions — Essential Hypertension; Heart Failure; Syncope; Dizziness; Hypertension

STUDY DESIGN:
Intervention Model Description: Intervention group: Participants in the intervention group were patients with hypertension who had been provided ADELE for the duration of the study. The observation period per participant was 3 months on average. Data on the primary, secondary and exploratory endpoints were gathered using questionnaires at study inclusion (t0) and an average of 3 months after randomization (t1). Control group: Participants in the control group were patients with hypertension who were not provided with ADELE for the duration of the study. The observation period per participant was 3 months on average. Data on the primary, secondary and exploratory endpoints were collected using questionnaires at study inclusion (t0) and an average of 3 months after randomization (t1).
  In addition, after the end of the observation period (from t0 to t1), the participants in the control group were offered an extension of a further 3 months on average using ADELE (from t1 to t2).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Participants in the intervention group were patients with hypertension who had been provided ADELE for the duration of the study. The observation period per participant was 3 months on average. Data on the primary, secondary and exploratory endpoints were gathered using questionnaires at study inclusion (t0) and an average of 3 months after randomization (t1).
  Interventions: Device: Digital health assistant ADELE
- Control group (No Intervention): Participants in the control group were patients with hypertension who were not provided with ADELE for the duration of the study. The observation period per participant was 3 months on average. Data on the primary, secondary and exploratory endpoints were collected using questionnaires at study inclusion (t0) and an average of 3 months after randomization (t1).
  In addition, after the end of the observation period (from t0 to t1), the participants in the control group were offered an extension of a further 3 months on average using ADELE (from t1 to t2).

INTERVENTIONS:
Device: Digital health assistant ADELE — The digital health assistant ADELE Blood Pressure A0007 (ADELE for short) improves the daily lives of patients with high blood pressure and enhances patient care. Participants in the intervention group were provided with ADELE to use during the study period for voice-based recording, interpretation and classification of their vital signs and body conditions.
  Arms: Intervention group

SUMMARY:
High blood pressure (hypertension) can cause damage to vital organs such as the heart, kidneys, eyes, brain and blood vessels. The risk of developing high blood pressure increases with age. High blood pressure is the leading risk factor for death worldwide. The digital health assistant ADELE Blood Pressure A0007 (ADELE for short) improves the daily lives of patients with high blood pressure and enhances patient care. The study aims to varify a positive effect of ADELE on the care of patients with hypertension. The study participants were randomly assigned to one of two groups. Participants in the intervention group were provided with ADELE to use during the study period for voice-based recording, interpretation and classification of their vital signs and body conditions. ADELE provides daily guideline-based knowledge modules on how to better manage the chronic disease. In addition, participants in the intervention group were able to use ADELE to set reminders, for example, to take their medication regularly, exercise regularly and drink enough. The participants in the control group were not provided with ADELE. The objective of the study is to prove a positive effect of the usage of ADELE on patient sovereignty, adherence (adherence to the therapy jointly agreed by patient and practitioner), health status, blood pressure values and health literacy in order to provide the basis for permanent admission to the routine care of the statutory health insurance if the effect is proven.

DETAILED DESCRIPTION:
Hypertension can cause damage to vital organs such as the heart, kidneys, eyes, brain and blood vessels. The risk of developing high blood pressure increases with age. Hypertension is the leading risk factor for death worldwide. The digital health assistant ADELE Blood Pressure A0007 (ADELE for short) improves the daily lives of patients with high blood pressure and enhances patient care. The study aims to varify a positive effect of ADELE on the care of patients with hypertension. The functions of ADELE are based on the recommendations of medical guidelines. The study was designed to confirm the positive care effect of the already empirically proven guideline recommendations in everyday use with ADELE.

A prospective randomized multicenter study with a parallel group design was used.

To conduct the study, adult participants with hypertension were randomly assigned to the intervention group or the control group as part of a 1:1 randomization. The observation period per participant was 3 months on average. The data was collected by means of questionnaires. ADELE was provided to the intervention group. ADELE was not provided to the participants in the control group. The primary objective of the study was defined as the improvement in patient sovereignty, measured after 3 months. The improvement in adherence, measured after 3 months, and the improvement in health status, measured after 3 months, were defined as secondary endpoints. The additional exploratory endpoints defined concern, for example, the reduction in systolic and diastolic blood pressure values and the improvement in health literacy.

The objective of the study is to prove a positive effect of the usage of ADELE on patient sovereignty, adherence (adherence to the therapy jointly agreed by patient and practitioner), health status, blood pressure values and health literacy in order to provide the basis for permanent admission to the routine care of the statutory health insurance if the effect is proven.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study
* Medically diagnosed and treated hypertension
* Regular use of at least 1 anti-hypertensive drug with increased overall cardiovascular risk or diabetes mellitus (stroke, heart attack, heart failure, CHD, after bypass / stent surgery, etc.) or 3 anti-hypertensive drugs
* Person must be able to understand the patient information
* Written informed consent form is signed at the beginning of interview 1

Exclusion Criteria:

* Persons belonging to specially protected groups (e.g. persons temporarily or permanently unable to give consent)
* Person suffers from mental illness that prevents them from understanding the information about the study, giving their consent or complying with the requirements of the study
* Person is unable to operate the application properly
* Person has already had contact with the application and/or a comparable application
* Person is participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Change of patient autonomy | From enrollment to the end of treatment at 3 months
  Change of patient autonomy, measured after 3 months based on Hypertension evaluation of lifestyle and management (HELM) scale. The HELM knowledge scale had 14 items across 3 domains: general hypertension knowledge, lifestyle and medication management, and measurement and treatment goals. The score is between 0 (Minimum) and 14 (Maximum). A higher value is better.

SECONDARY OUTCOMES:
Change of adherence | From enrollment to the end of treatment at 3 months
  Change of adherence, measured after 3 months based on Hill-Bone Compliance to High Blood Pressure Therapy Scale (HB-HBP). The scale is based on 14 items. Minimum is 56, Maximum is 0. A lower score is better.
Change of health condition | From enrollment to the end of treatment at 3 months
  Change of health condition, measured after 3 months using Short Form 12 Health Survey (SF-12). The scale is based on 12 items. The score is between 0 (Minimum) and 100 (Maximum). A higher value is better.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hoffmann, Prof. Dr. med., Study Chair — (Minority) shareholder; Oliver Vonend, Prof. Dr. med., Principal Investigator — No affiliation; Hans-Peter Reiffen, Prof. Dr. med., Study Director — No affiliation
Locations (2):
- Germany (2):
  - Ökumenische Sozialstation Heidenheimer Land, Heidenheim, Baden-Wurttemberg
  - Johanniter-Unfall-Hilfe e.V., Hanover, Lower Saxony

IPD SHARING:
Plan to Share IPD: No